CLINICAL TRIAL: NCT04798677
Title: Efficacy and Tolerability of a Nutritional Supplementation With ABBC-1, a Symbiotic Combination of Beta-glucans and Selenium and Zinc Enriched Probiotics, in Volunteers Receiving the Influenza or the Covid-19 Vaccines
Brief Title: Efficacy and Tolerability of ABBC1 in Volunteers Receiving the Influenza or Covid-19 Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: HMDM/ABBC-1/v4
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Immunity; Vaccine Reaction; Influenza; Covid19; Cytokine Storm; Immunologic Deficiency Syndromes
Keywords: Trained immunity; Vaccine adjuvant; Influenza; Covid-19; beta-glucans; Saccharomyces cerevisiae; microbiota; ABBC1
MeSH Terms: conditions — Influenza, Human; COVID-19; Cytokine Release Syndrome; Immunologic Deficiency Syndromes

STUDY DESIGN:
Intervention Model Description: Single-center, randomized, double-blinded, placebo-controlled clinical study. Multicomponent intervention (clinical and nutritional) resulting from the administration of influenza or Covid-19 vaccine and supplementation with ABBC-1.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Ramdomized, double-blinded and placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Influenza vaccine + intervention with beta-glucan complex and Saccharomyces cerevisiae consortium (Experimental): Influenza vaccine followed by 30 days of supplementation with a beta-glucan complex and Saccharomyces consortium rich in selenium and zinc
  Interventions: Dietary Supplement: ABBC1 Immunoessential
- Influenza vaccine + placebo (Placebo Comparator): Influenza vaccine followed by 30 days of supplementation with a placebo, similar en aspect, flavor and odour to the intervention product
  Interventions: Dietary Supplement: Placebo
- Covid-19 vaccine + intervention with beta-glucan complex and Saccharomyces cerevisiae consortium (Experimental): Covid-19 vaccine followed by 35 days of supplementation with a beta-glucan complex and Saccharomyces consortium rich in selenium and zinc
  Interventions: Dietary Supplement: ABBC1 Immunoessential
- Covid-19 vaccine + placebo (Placebo Comparator): Covid-19 vaccine followed by 30 days of supplementation with a placebo, similar en aspect, flavor and odour to the intervention product
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ABBC1 Immunoessential — Powder for dissolution in water, based on a yeast beta-glucan complex and a consortium of Saccharomyces cerevisiae rich in selenium and zinc + excipents. Lemon flavor
  Arms: Covid-19 vaccine + intervention with beta-glucan complex and Saccharomyces cerevisiae consortium; Influenza vaccine + intervention with beta-glucan complex and Saccharomyces cerevisiae consortium
Dietary Supplement: Placebo — Powder for dissolution in water, excipents. Lemon flavor
  Arms: Covid-19 vaccine + placebo; Influenza vaccine + placebo

SUMMARY:
The immune system response needs to be forceful but also balanced for a rapid recovery from infection which avoids harmful overreactions. Innate immunity can adapt and respond more efficiently to secondary exposures, thanks to epigenetic and metabolic reprogramming, namely "trained immunity".

ABBC1 is a combination of beta-1,3/1,6-glucan with inactivated Saccharomyces cerevisae rich in selenium and zinc for training immunity. ABBC1 includes repurposed synergistic yeast-based ingredients: a unique ß-1,3/1,6-glucan complex and a consortium of probiotic Saccharomyces cerevisiae, rich in Selenium and Zinc. ABBC1 induces trained immunity due to its specific chemical and tridimensional structure: its ß-glucan complex interacts with specific receptors in immune cells, provoking a release of cytokines and priming phagocytosis. Simultaneous activation of these pathways activates innate immunity and counteracts cytokine storm.

ABBC1 provides highly bioavailable selenium and zinc, micronutrients with a critical role in an optimal immune responsiveness to allergy, infection, and vaccines. ABBC1 possesses proven microbiome modulating properties, which revert in immune training. Due to its high tolerance, safety and immediate availability, ABBC1 is an ideal candidate for complementary management of geriatric patients with seasonal influenza viruses or COVID-19, or to improve the immune response in the general population receiving the influenza or Covid-19 vaccines. The absence of drug interactions in ABBC1 allows a dosage that is fully compatible with the medication prescribed for all types of patients, including the elderly who are frequently polymedicated, and allows adding an additional therapeutic tool in the fight against the pandemic.

This study assesses the benefits of a nutritional supplementation with ABBC1 in volunteers receiving the influenza vaccine during autumn 2020 and the Covid-10 vaccine during winter 2021.

DETAILED DESCRIPTION:
On March 11, 2020, the World Health Organization (WHO) declared the COVID-19 disease caused by SARS-CoV-2 (Severe Acute Respiratory Syndrome Coronavirus 2) as a pandemic. The Covid-19 pandemic is evolving throughout the world and is associated with high mortality and morbidity. According to Salem ML et al. 2020, the influenza vaccine may have an adjuvant effect to minimize the severity of COVID-19, since the correlation of Covid-19-related mortality and morbidity and the influenza vaccination situation appears to be protective. The trend of the correlation could be explained in parameters of incidence and recovery of cases.

Vaccination against influenza (H1N1) is cost-effective and safe. Given that the influenza virus shares some common epitopes and mechanisms with the SARS-CoV-2 virus, there is the possibility of partial protection for reduce severity related to Covid-19 through flu vaccination. The influenza viruses and the SARS-CoV-2 viruses have an evolutionary proximity. Since this vaccination is not mandatory for routine clinical practice, various countries adopt different policies, and vaccination rates differ considerably among them. For this reason, the WHO in February 2020 published a recommendation on the composition of vaccines against influenza virus for use in the 2020-2021 northern hemisphere influenza season.

Under this situation, it has been identified that older adults and people suffering from serious chronic conditions such as heart disease, lung disease or kidney disease have a higher risk of suffering from severe COVID-19. Older people are twice as likely to have severe COVID-19. This is probably because as people age, their immune systems change, making it harder to fight off disease and infection, and for this reason age is considered a risk factor for the disease.

After several months of the global impact of the pandemic, specific vaccines for Covid-19 will begin to be available by end 2020. In Spain, the Ministry of Health designed a vaccination plan that will begin immediately. Specifically, in Catalonia this plan foresees classifying the population into various risk groups, based on highest priority and immediacy. Older adults make up one of the groups that will receive the vaccine as a priority. At the same time, they represent a population group whose immune response after the administration of other vaccines has been found to be less effective or optimal than in healthy adults under 65 years of age. For example, the influenza vaccine has an efficacy of 70-90% in the general population, while this efficacy is reduced to 17-53% in adults older than 65 years. In the same line, preliminary results with Covid-19 vaccines observe a better efficacy (> 90%) in groups of people under 55 years of age compared to those over 55 years of age (62%), results that suggest that the efficacy could decrease with age.

The reduced efficacy of vaccines in the elderly may be because the geriatric population frequently presents immunosenescence (or a decline in immune function due to aging), but also to a possible poor nutritional status, in which it is not achieved to reach an optimal supply of essential oligonutrients for an effective antiviral immune response.

Specifically, the efficacy data for the BNT162b2 vaccine in people older than 65 years considered a risk population point to a slightly lower efficacy (91.7% versus 94.8% in the general population). However, the results point to less protection after the administration of a single dose of the vaccine (82.0% efficacy just after the administration of the first dose and 52.4% between doses 1 and 2, compared to 94.8% 7 Days after the second dose), regardless of age. This requires a long administration schedule that does not make protection effective until a month after the first administration, slowing down access to the vaccine to a greater part of the population and leaving around 18-48% of unprotected vaccinated population until the administration of the second dose. The benefits of increasing efficacy after the first dose could be of great importance for Public Health since it would allow a more immediate immunization of the vaccinated population even before the administration of the second dose.

A higher and faster immune response to the vaccine could benefit not only the elderly population, but also any other type of sub-population to be vaccinated. The group of medical staff workers represents a population subject to constant exposure to the virus, and for this reason it is considered another priority group to receive the vaccine. This group will be exposed to infection during the window of time that passes between the administration of the first and the second dose, so the possibility of improving the immune response immediately could have a huge benefit.

Over the past 10 years, a wide range of pleiotropic effects of selenium have been discovered, ranging from antioxidant and anti-inflammatory effects to the production of active thyroid hormone, which has drawn attention to the relevance of selenoproteins for health. Low selenium level has been associated with an increased risk of mortality, poor immune function, and cognitive decline. An increased level of selenium or selenium supplementation has antiviral effects, is essential for the success of male and female reproduction and reduces the risk of autoimmune thyroid diseases. Older adults with insufficient selenium intake are at increased risk for a poorer clinical outcome after viral exposure due to a response sub-optimal antiviral response. Results from an intervention clinical trials have shown that daily supplementation of older adults with 100 ug of high selenium yeast can raise plasma selenium levels to 150 ug / L, which is within the proposed target range of selenium status. High selenium yeast has demonstrated its safety and clinical efficacy in human supplementation trials.

On the other hand, the low to moderate zinc deficiency that is highly prevalent in elderly persons mimics many of the features of the immunosenescence of aging. Therefore, some of the deficits in immune regulation seen among the elderly could be ameliorated or reversed through daily zinc supplementation. It has been demonstrated that low zinc status is associated with increased risk of respiratory disease, including pneumonia, and inflammation. Research indicates that zinc supplementation can restore serum zinc levels in some elderly persons with low zinc status. Zinc supplementation of 15 per day that may increase immune readiness and favor regulated immune response. This protective approach may be particularly important in individuals who may be prone to cytokine-driven immune overreaction during the COVID-19 epidemic.

Finally, the immunostimulatory effect of beta-glucan is widely known. Specifically, yeast or fungal beta-1,3/1,6-glucans interact with specific receptors (dectin-1, TLR2 and 6 or CR3) in different cells of the immune system, such as macrophages, neutrophils, granulocytes, Natural Killer cells or dendritic cells. This interaction stimulates the production of antibodies and primes phagocytosis, strengthening defense mechanisms against infections. It is important to note that not all beta-glucans have the same mechanisms of action: while other linear beta-glucans only bind to Dectin-1 and promote a reduction of phagocytosis and cytokine secretion, beta-1,3/1,6-glucans, branched polymers that simultaneously stimulate Dectin-1 and TLR4 receptors, stimulate phagocytosis, activate innate immunity and prevent or counteract exacerbated immune reactions, allergy or inflammation. In addition, these effects are improved in combination with selenium.

ABBC1 is a combination of beta-1,3/1,6-glucan with inactivated Saccharomyces cerevisae rich in selenium and zinc for immunity enhancement. Due to its high tolerance, safety and immediate availability, ABBC1 is an ideal candidate for complementary management for geriatric patients with seasonal influenza viruses or COVID-19, or to improve the immune response in the general population receiving the influenza or Covid-19 vaccines. The absence of drug interactions in ABBC1 allows a dosage that is fully compatible with the medication prescribed for all types of patients, including the elderly who are frequently polymedicated, and allows adding an additional therapeutic tool in the fight against the pandemic.

In this study we propose to determine the benefits of supplementation with ABBC1 in volunteers receiving the influenza vaccine at a first stage and the Covid-19 vaccine when available, to study if their immune response to the vaccine improves and/or leads to a better clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

COMMON CRITERIA:

* Subjects with the ability to take the study product orally
* Ability to understand the study, the information about the symptoms and to comply with the treatment shots.
* Subject or legal guardian / representative willing to give informed consent in writing.

INFLUENZA VACCINE GROUPS:

* Subjects who require hospitalization or external follow-up (outpatients or PADES)
* Subjects over 60 years old who will receive the influenza vaccine

COVID-19 VACCINE GROUPS

* Subjects from long-stay centres attached to the Hospital Mare de Déu de la Mercè, and meet the following inclusion criteria:
* Groups:

  * Subjects over 18 years of age who receive the Covid-19 vaccine, in a stable clinical situation, at the discretion of the researcher, or
  * Healthcare workers of the study centers, over 18 years of age who receive the Covid-19 vaccine
* Availability to attend clinical visits.

Exclusion Criteria:

COMMON CRITERIA:

* Need for assisted ventilation that makes oral consumption of the product under study impossible
* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active principle or to any of the excipients.
* History or evidence of any medical conditions or medication use that, in the opinion of the principal investigator, could affect the safety of the subjects or interfere with the study evaluations
* Subjects in situation of last days

COVID-19 VACCINE GROUPS:

* Subjects in whom the Covid-19 vaccine is contraindicated.
* A history of frailty or comorbidity that indicates a situation of clinical instability.
* History or evidence of any medical conditions or drug use that, in the opinion of the principal investigator, could affect the safety of subjects or interfere with study evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-09-24 (Actual)

PRIMARY OUTCOMES:
Change in the acute immune response to the influenza vaccine after supplementation (influenza vaccine groups) | 30 days (Days 1, 7 and 30)
  Generation of T-cells (TCD8, TCD3 and TCCD4)
Change in the delayed immune response to the influenza vaccine after supplementation (influenza vaccine groups) | 30 days (Days 1, 7 and 30)
  Generation of influenza-specific antibodies (IgM, IgG influenza A and B)
Change in the acute immune response to the Covid-19 vaccine after supplementation (Covid-19 vaccine groups) | 35 days (Days 1, 7, 21 and 35)
  Generation of T-cells (TCD8, TCD3 and TCCD4)
Change in the delayed immune response to the Covid-19 vaccine after supplementation (Covid-19 vaccine groups) | 35 days (Days 1, 7, 21 and 35)
  Generation of influenza-specific antibodies (IgM, IgG influenza A and B)
Change in blood levels of selenium and zinc | 30 days (Days 1, 7 and 30) for influenza vaccine groups. 35 days (Days 1, 7, 21 and 35) for Covi-19 groups.
  Variation of selenium and zinc levels measured in plasma

SECONDARY OUTCOMES:
Incidence of influenza (only for influenza vaccine groups) | 30 days
  Number of volunteers presenting influenza as measured by clinical diagnostic
Incidence of Covid-19 | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Number of volunteers presenting Covid-19 as measured by clinical diagnostic and/or PCR or antigen test
Mean Change in the Ordinal Scale WHO R&D Blueprint novel Coronavirus | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. A positive change indicates a worsening and a negative change is an improvement.
Number of subjects with fever during the study | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Variation on body temperature (ºC)
Number of subjects with cough during the study | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Clinical assessment
Number of subjects with myalgia during the study | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Clinical assessment
Number of subjects with dyspnea during the study | 30 days for influenza groups, 35 days for Covid-19 groups
  Clinical assessment
Number of subjects with anosmia / ageusia during the study | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Clinical assessment
Hospital readmission rate during the study and the additional follow-up period | 60 days
  percentage of patients readmitted to the hospital during the study and the addition follow-up period
Changes in blood glucose | 30 days for influenza groups, 35 days for Covid-19 groups
  measured in blood samples
Incidence of adverse effects of the study product | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  reporting of adverse events (if any)
Dietary history | 30 days for influenza vaccine groups, 35 days for Covid-19 vaccine groups
  Record of the dietary history during the study

OTHER OUTCOMES:
Blood analysis (Influenza vaccine groups) | 30 days
  Alterations in the blood count and in inflammatory or immune function markers
Blood analysis (Covid-19 vaccine groups) | 35 days
  Alterations in the blood count and in inflammatory or immune function markers

CONTACTS AND LOCATIONS:
Overall Officials: Julián A. Mateus Rodríguez, MD, PhD, Principal Investigator — Hospital Mare de Deu de la Mercè - Germanes Hositalàries
Locations (1):
- Hospital Mare de Déu de la Mercè - Germanes Hospitalàries, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
IPD will be available upon request (blood analysis results and clinical assessment outcomes)

REFERENCES:
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Knoll MD, Wonodi C. Oxford-AstraZeneca COVID-19 vaccine efficacy. Lancet. 2021 Jan 9;397(10269):72-74. doi: 10.1016/S0140-6736(20)32623-4. Epub 2020 Dec 8. No abstract available. PMID 33306990
- [Result] Salem ML, El-Hennawy D. The possible beneficial adjuvant effect of influenza vaccine to minimize the severity of COVID-19. Med Hypotheses. 2020 Jul;140:109752. doi: 10.1016/j.mehy.2020.109752. Epub 2020 Apr 22. No abstract available. PMID 32361099
- [Result] Arokiaraj MC. Considering Interim Interventions to Control COVID-19 Associated Morbidity and Mortality-Perspectives. Front Public Health. 2020 Sep 22;8:444. doi: 10.3389/fpubh.2020.00444. eCollection 2020. PMID 33072682
- [Result] Menachery VD, Debbink K, Baric RS. Coronavirus non-structural protein 16: evasion, attenuation, and possible treatments. Virus Res. 2014 Dec 19;194:191-9. doi: 10.1016/j.virusres.2014.09.009. Epub 2014 Sep 30. PMID 25278144
- [Result] Zeng Q, Langereis MA, van Vliet AL, Huizinga EG, de Groot RJ. Structure of coronavirus hemagglutinin-esterase offers insight into corona and influenza virus evolution. Proc Natl Acad Sci U S A. 2008 Jul 1;105(26):9065-9. doi: 10.1073/pnas.0800502105. Epub 2008 Jun 11. PMID 18550812
- [Result] Wang J, Tang K, Feng K, Lin X, Lv W, Chen K, Wang F. Impact of temperature and relative humidity on the transmission of COVID-19: a modelling study in China and the United States. BMJ Open. 2021 Feb 17;11(2):e043863. doi: 10.1136/bmjopen-2020-043863. PMID 33597143
- [Result] Rayman MP. Selenium and human health. Lancet. 2012 Mar 31;379(9822):1256-68. doi: 10.1016/S0140-6736(11)61452-9. Epub 2012 Feb 29. PMID 22381456
- [Result] Goldson AJ, Fairweather-Tait SJ, Armah CN, Bao Y, Broadley MR, Dainty JR, Furniss C, Hart DJ, Teucher B, Hurst R. Effects of selenium supplementation on selenoprotein gene expression and response to influenza vaccine challenge: a randomised controlled trial. PLoS One. 2011 Mar 21;6(3):e14771. doi: 10.1371/journal.pone.0014771. PMID 21445287
- [Result] Prasad AS, Beck FW, Bao B, Fitzgerald JT, Snell DC, Steinberg JD, Cardozo LJ. Zinc supplementation decreases incidence of infections in the elderly: effect of zinc on generation of cytokines and oxidative stress. Am J Clin Nutr. 2007 Mar;85(3):837-44. doi: 10.1093/ajcn/85.3.837. PMID 17344507
- [Result] Meydani SN, Barnett JB, Dallal GE, Fine BC, Jacques PF, Leka LS, Hamer DH. Serum zinc and pneumonia in nursing home elderly. Am J Clin Nutr. 2007 Oct;86(4):1167-73. doi: 10.1093/ajcn/86.4.1167. PMID 17921398
- [Result] Barnett JB, Dao MC, Hamer DH, Kandel R, Brandeis G, Wu D, Dallal GE, Jacques PF, Schreiber R, Kong E, Meydani SN. Effect of zinc supplementation on serum zinc concentration and T cell proliferation in nursing home elderly: a randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2016 Mar;103(3):942-51. doi: 10.3945/ajcn.115.115188. Epub 2016 Jan 27. PMID 26817502
- [Result] Vetvicka V, Vannucci L, Sima P, Richter J. Beta Glucan: Supplement or Drug? From Laboratory to Clinical Trials. Molecules. 2019 Mar 30;24(7):1251. doi: 10.3390/molecules24071251. PMID 30935016
- [Result] Engstad RE, Robertsen B. Recognition of yeast cell wall glucan by Atlantic salmon (Salmo salar L.) macrophages. Dev Comp Immunol. 1993 Jul-Aug;17(4):319-30. doi: 10.1016/0145-305x(93)90004-a. PMID 8375567
- [Result] Raa J. Immune modulation by non-digestible and non-absorbable beta-1,3/1,6-glucan. Microb Ecol Health Dis. 2015 May 29;26:27824. doi: 10.3402/mehd.v26.27824. eCollection 2015. No abstract available. PMID 26031679
- [Result] Vetvicka V, Vannucci L, Sima P. beta-glucan as a new tool in vaccine development. Scand J Immunol. 2020 Feb;91(2):e12833. doi: 10.1111/sji.12833. Epub 2019 Nov 13. PMID 31544248
- [Result] Novak M, Vetvicka V. Glucans as biological response modifiers. Endocr Metab Immune Disord Drug Targets. 2009 Mar;9(1):67-75. doi: 10.2174/187153009787582423. PMID 19275682
- [Result] De Marco Castro E, Calder PC, Roche HM. beta-1,3/1,6-Glucans and Immunity: State of the Art and Future Directions. Mol Nutr Food Res. 2021 Jan;65(1):e1901071. doi: 10.1002/mnfr.201901071. Epub 2020 Apr 27. PMID 32223047
- [Result] Fulop T, Dupuis G, Witkowski JM, Larbi A. The Role of Immunosenescence in the Development of Age-Related Diseases. Rev Invest Clin. 2016 Mar-Apr;68(2):84-91. PMID 27103044
- [Result] Goodwin K, Viboud C, Simonsen L. Antibody response to influenza vaccination in the elderly: a quantitative review. Vaccine. 2006 Feb 20;24(8):1159-69. doi: 10.1016/j.vaccine.2005.08.105. Epub 2005 Sep 19. PMID 16213065
- [Result] Polack FP, Thomas SJ, Kitchin N, Absalon J, Gurtman A, Lockhart S, Perez JL, Perez Marc G, Moreira ED, Zerbini C, Bailey R, Swanson KA, Roychoudhury S, Koury K, Li P, Kalina WV, Cooper D, Frenck RW Jr, Hammitt LL, Tureci O, Nell H, Schaefer A, Unal S, Tresnan DB, Mather S, Dormitzer PR, Sahin U, Jansen KU, Gruber WC; C4591001 Clinical Trial Group. Safety and Efficacy of the BNT162b2 mRNA Covid-19 Vaccine. N Engl J Med. 2020 Dec 31;383(27):2603-2615. doi: 10.1056/NEJMoa2034577. Epub 2020 Dec 10. PMID 33301246